CLINICAL TRIAL: NCT04692441
Title: APOE Genotype Effects on Triglycerides and Blood Flow in the Human Brain
Brief Title: Apolipoprotein E (APOE) Genotype Effects on Triglycerides and Blood Flow in the Human Brain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Angela Hanson, Assistant Professor, School of Medicine, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00009772; 1R01AG067563-01 (NIH)
Record Dates: First submitted 2020-11-19; First posted 2020-12-31 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Alzheimer Disease; Dementia
Keywords: APOE genotype; lipid metabolism
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Intervention Model Description: Each participant undergoes the same intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): All participants undergo the same intervention: Drinking heavy cream and undergoing MRI.
  Interventions: Dietary Supplement: Heavy Cream

INTERVENTIONS:
Dietary Supplement: Heavy Cream — 100 ml of dairy cream with 40.4g of total fat, to ingest orally

SUMMARY:
High fat feeding (HFF) increases the risk of Alzheimer's disease (AD) but individuals who carry the AD risk gene E4 paradoxically improve after acute HFF. The investigators propose to further study this phenomenon with a clinical study to assess cerebral blood flow which can be measured by a technique called arterial spin labeling (ASL) on an MRI and is tightly related to brain metabolism.

DETAILED DESCRIPTION:
Overview: The purpose of the study is to enroll 90 older adults, half of whom will have E4 carrier status, to assess whether E4 status affects change in global cerebral blood flow (∆CBF) in response to a high fat drink. The screening visit includes informed consent, baseline blood draw, oral triglyceride tolerance test (OTTT), and dual-energy x-ray absorptiometry (DEXA). The study visit involves assessing cerebral blood flow using arterial spin labeling (ASL) MRI - at baseline and at 2 hours after drinking heavy cream. The study visit will also include 6 blood draws and a 30 minute cognitive battery.

Screening Visit Procedures (at Seattle South Lake Union campus): Before the screening visit, participants will receive a copy of the consent form in the mail as well as a medical history questionnaire to fill out. Participants will be advised to fast the night before the screening visit (minimum 8 hours required). After an informed consent process, study personnel will check vitals, including waist circumference, height, and weight for body mass index (BMI) calculation. An IV will be placed by the study nurse and blood sent for complete blood count, chem20 (including liver and kidney function assessment), glycated hemoglobin (hemoglobin A1C), lipid panel, and a blood sample for APOE genotyping (Northwest Lipids using polymerase chain reaction (PCR) methodology). Blood samples except APOE will be sent to the University of Washington (UW) Clinical Laboratory Improvement Amendment (CLIA)-certified lab, and participants will receive a copy of the results by mail. After the blood draw, participants will then undergo an oral glucose tolerance test (OGTT): 6 time points (0, 15, 30, 45, 60,120 min) which will include a blood draw for plasma to measure insulin and C peptide (in batches by Northwest (NW) lipids). At time 0 and 120 minutes study personnel will also assess vitals and a point of care glucose using a glucometer. The OGTT will be the standard 75 grams glucose drink from central supply. After the 2-hour OGTT is complete, patients will undergo a DEXA scan. Note, DEXA can be performed before OGTT if needed for study flow. Parking will be provided, and participants will be paid with a gift card.

Screening visit sample day:

8 am: Check in to the clinic 8-8:30: informed consent in private room, go over medical history 8:30-9: Insert IV, fill out depression, anxiety screen, draw baseline blood 9 -11 am: OGTT (During gaps in OGTT, do Montreal Cognitive Assessment (MoCA)) 11-11:25 am: DEXA 11:25-11:30: Remove IV, distribute gift card and parking validation Time: 3.5 hours, total blood drawn 40 mls

Study Visit Procedures (at University of Washington main campus): Participants will arrive to the UW Translational Research Unit (TRU) after an overnight fast (minimum 8 hours required). The study nurse will place an IV, and check vital signs including blood pressure, heart rate, temperature, and weight. Then, the participant will be escorted to the MRI scanner and undergo the fasting imaging protocol. The participant will head back to the TRU and start the oral triglyceride tolerance test (OTTT). Time 0 blood is drawn and time documented. Then, the participant will drink the dairy product-100 mLs of heavy cream (just under half a cup) which contains 370 calories, 40.4 grams of total fat, 23.6 grams of saturated fat. The participant will be encouraged to drink the product over 5 minutes as per published OTTT protocols. Blood draws will be collected for measurement of glucose, insulin, lipids and appetite hormones (30, 120, 180, 240 min). A post-lipid MRI will be done at the 2 hour time point, and the NIH toolbox cognitive assessment will be done at 3 hour time point. The NIH battery takes approximately 30 minutes to administer and will be done on a portable tablet.

Study visit sample day:

8 am: Check in to UW TRU, ask about new medications, place IV 8:15: Escort down to MRI area, get pre-MRI 8:45: Back at TRU: T0 blood draw 8:45-8:50: Drink lipid 9:20: T30 min blood draw 9:50: T60 min blood draw 10:50: T120 min (2 hour) blood draw

**Return to MRI scanner for 2 hour MRI** (will be ~2 hours and 10 minutes post drink) 11:50: T180 min (3 hour) blood draw **Do the NIH toolbox testing now - takes about 30 minutes** 12:50: T240 min (4 hour) blood draw 12:50-1 pm: Remove IV, receipt of gift card, participant checks out. Time: 5 hours, total blood drawn: 80 mls (13 per blood draw x 6 time points)

MRI protocol: The investigator will use pseudo-continuous arterial spin labeling to measure cerebral blood flow (CBF) in ml/100g/min as a marker of perfusion for improved signal quality. In this approach, magnetically labeled arterial blood water serves as the endogenous contrast. MRI images will be stored on external hard drive with encryption and will be uploaded to One Drive or another HIPAA-compliant system for further processing and analysis.

Experiment: As per the consensus recommendations, the investigator will use a sequence (5.5 minutes) with long label duration = 1.8 s, long post-labeling delay = 2 s, with labeling offset = 25-30 mm, slices = 20, spatial resolution = 3.5×3.5×5 mm3, field of view = 240×240×100 mm3, SENSE-factor = 2, repetition time/echo time (TR/TE)= 5000/18 ms. Dual adiabatic background suppression pulses will be applied to minimize gray and white matter tissue contamination at inversion delay (TI) = 2.05 and 3.25 s. Finally, the investigator will acquire an equilibrium magnetization scan (M0, 1 minute), identical to the above scan, but with TR = 10,000 ms and no labeling or background suppression.

Analysis: First, motion correction will be applied to the arterial spin labeling images using motion correction (FSL-MCFLIRT), and these will be registered to the M0 image. Then, the investigator will perform a pair-wise subtraction between the control and null images and apply a two-compartment model to quantify CBF. The resulting CBF map will be co-registered to the T1 scan followed by a transformation to Montreal Neurological Institute (MNI) space.The temporal regions such as the entorhinal cortex, temporal lobe, hippocampus as well as the posterior cingulate and lateral parietal lobules will be identified using standard Harvard-Oxford Cortical and Subcortical atlas. CBF values will be compared in these regions between the groups. The region of interest approach can dilute effects that are smaller than the size of the region of interest. Therefore, the investigator will also perform permutations testing in FSL to evaluate voxel-wise CBF differences between group. In order to ensure that the voxel-wise outcomes are not mere chance, the investigator will impose strict family-wise error correction for multiple comparisons.

Data collected for this study:

Data collected on the phone and on medical history form (verbal consent given, prior to informed consent):

Medical history, including if participants know their APOE genotype Targeted review of systems Age of menopause (for women) Medications Use of drugs, tobacco, and alcohol Drug allergies Food allergies/intolerances Handedness Work and Education history of participant Education level of mother (if known) Education level of father (if known) MRI checklist: surgeries, metal in body

Data collected at screening visit:

How patient identifies as to race/ethnicity Vitals: Height, weight, waist circumference measures Physical Health Questionnaire-9 (PHQ9, a depression screen) Generalized Anxiety Disorder-7 Assessment (GAD-7, an anxiety screen) Cognitive assessment: MoCA version 8.2 English version Screening bloodwork: chemistries, hepatic function, lipid panel, hemoglobin A1C, Complete Blood Count (CBC), APOE genotype (cheek swab and blood test) Fasting and 2 hour point of care glucose (using a glucometer) Fasting and 2 hour heart rate, blood pressure Six OGTT blood draws: 4 ml lavender top tube to measure glucose, insulin (sent to lab in batches) DEXA scan for standard body composition measures (i.e. fat mass, fat-free mass)

Data collected at study visit:

Vitals: Heart Rate (HR), BP, Respiratory Rate (RR), temperature at all time points Six blood draws: serum and plasma collection for glucose, insulin, lipids and appetite hormones NIH toolbox cognitive data MRI ASL data: Total and regional ASL images (does not include a clinical MRI read)

ELIGIBILITY:
Inclusion Criteria:

1. Aged 55 or older at the date of the screening visit
2. Equal representation of APOE E4 carriers and non-carriers
3. Strive for equal numbers of men and women; women need to be post-menopausal for at least 1 year or medical equivalent (hysterectomy)
4. Able to read and understand English
5. Able to cognitively and physically give informed consent 6.Able to undergo an MRI and ingest dairy products

Exclusion Criteria:

1. Diabetes requiring medication: Known type 1 or type 2 diabetes requiring oral diabetic medications or insulin. Diet-controlled diabetes, 'pre-diabetes,' remote use of diabetic agents, or a history of gestational diabetes is ok to enroll.
2. Hypertension requiring medication: Participants taking medication for hypertension will be excluded, unless they can safely stop the medication for 2 weeks, per their primary care provider, before the study visit (The MRI visit).
3. Significant lipid abnormalities: Diagnosis of hyperlipidemia requiring statin, bile acid resins, fibrate medications, and/or high dose niacin will be excluded. If participants are willing to stop their medications 4 weeks before the screening visit (as long as they are not on medication for secondary prevention of heart attack or stroke), this is ok. If participants are taking over-the-counter medications known to affect lipid metabolism including omega-3 fatty acids, niacin, or red yeast rice, they can enroll if they agree to stop the medication 4 weeks before the screening visit. Also excluded are significant cholesterol abnormalities as defined by the 2018 American College of Cardiology/American Heart Association (ACC/AHA) lipid guidelines including a fasting LDL cholesterol ≥190 mg/dL or fasting triglycerides > 500 mg/dL. Total cholesterol levels and HDL levels outside of the typical range are ok.
4. Dementia and cognitive impairment: Known diagnosis of dementia, use of dementia medications, or identification of dementia during the baseline visit, will be excluded. Also excluded are other significant neurologic diseases which affect cognition, such as recent stroke, recent severe head injury, or advanced Parkinson's disease. Mild cognitive impairment with no functional deficits is ok.
5. Psychiatric disorders: Participants who report active untreated major depression, psychosis, or mania, or who present with those symptoms at the baseline visit, or who act belligerent or unprofessional toward the clinical staff, will be excluded. Psychiatric conditions which are stable and treated with medication or therapy are ok. Similarly, individuals who meet criteria for active alcohol or drug abuse disorder will also be excluded as many of these substances could affect the study outcome.
6. Other significant medical illnesses: Illnesses which would cause a hardship on the participant to attend study visits and undergo a glucose tolerance test and an MRI. This includes unstable angina, moderate or severe chronic obstructive pulmonary disease (COPD), class III-IV Congestive heart failure (CHF), active liver or kidney disease causing cognitive symptoms, active cancer undergoing systemic chemotherapy or radiation, as well as other illnesses which in the study physician's view would put the participant at risk and also may place an undue burden on the participant.
7. Major digestive disorders: Disorders which would affect fat tolerance and absorption will be excluded including inflammatory bowel disease, gastric bypass or banding, or small intestine resection. Also excluded are allergies or major intolerance to milk or dairy products.
8. Contraindications to MRI: Metal in body that is not compatible with an MRI, other conditions that preclude an MRI (such as not being able to lie still or lie flat for an extended time) are excluded.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in global cerebral blood flow between baseline and 2 hours post lipid ingestion (Change CBF) | 2 Hour Change
  Change in global cerebral blood flow (CBF) in ml/100g/min, calculated as the subtracted difference between the pre- and the post-ASL flow in response to the intervention.

SECONDARY OUTCOMES:
Change in regional CBF | 2 Hour Change
  Change in regional cerebral blood flow (standard brain regions identified using standard Harvard-Oxford Cortical and Subcortical atlas) in ml/100g/ min, calculated as the difference between the pre- and the post-ASL flow in response to the intervention.
Fluid Cognitive Composite Standard Score | 3 hours post-drink ingestion
  The fluid cognitive composite standard score, from the National Institute of Health Toolbox cognitive assessment. Scores are expressed as normalized averages. Scores range from 0 to 140; a score of 100 represents an average ability, and higher scores indicate an above-average ability.

OTHER OUTCOMES:
Change in global cerebral blood flow as correlated with exploratory factors | 2 Hour Change
  Exploratory factors include fasting lipid levels, fasting and 2 hour OGTT glucose levels, hemoglobin A1C, and fat mass as assessed by DEXA.
Change in regional cerebral blood flow as correlated with exploratory factors | 2 Hour Change
  Exploratory factors include fasting lipid levels, fasting and 2 hour OGTT glucose levels, hemoglobin A1C, and fat mass as assessed by DEXA.

CONTACTS AND LOCATIONS:
Overall Officials: Angela J Hanson, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No